CLINICAL TRIAL: NCT01872741
Title: Prospective Randomized Study Comparing Clinical, Functional and Aesthetics Results of "Classical" Pterional and Minipterional Craniotomies.
Brief Title: Minipterional Versus Pterional Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Leonardo C. Welling, MD, Post graduation programm, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MiniPT Trial
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Intracranial Aneurysm; Muscular Atrophy
Keywords: craniotomy,; intracerebral aneurysms,; atrophy,; temporal muscle,; outcome
MeSH Terms: conditions — Intracranial Aneurysm; Muscular Atrophy; Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ruptured intracranial aneurysms (Active Comparator): Pterional craniotomy Minipterional craniotomy
  Interventions: Procedure: Minipterional craniotomy; Procedure: Pterional craniotomy
- Unruptured intracranial aneurysms (Active Comparator): Pterional craniotomy Minipterional craniotomy
  Interventions: Procedure: Minipterional craniotomy; Procedure: Pterional craniotomy

INTERVENTIONS:
Procedure: Minipterional craniotomy — Minipterional craniotomy approach for ruptured and unruptured aneurysms
Procedure: Pterional craniotomy — Pterional craniotomy approach for ruptured and unruptured aneurysm

SUMMARY:
This randomized prospective study was designed to compare the clinical, functional and aesthetic results of two surgical techniques for microsurgical clipping of anterior circulation aneurysms

DETAILED DESCRIPTION:
This randomized prospective study was designed to compare the clinical, functional and aesthetic results of two surgical techniques for microsurgical clipping of anterior circulation aneurysms. Overall, 60 eligible patients admitted with ruptured and unruptured anterior circulation aneurysms will enrolled in the study.

The aesthetic results will be analyzed with 2 methods. In the first, the patients will be showed to a rule, with a scale from 0 to 100, in which 0 mean the best result and 100 the worst result. Photos will be taken and showed to two independent observers, the results will be classified as excellent, good, regular or poor. The degree of atrophy will be measured with three methods. In the first one, the authors wiil observes the percentage of thick reduction in the temporal muscle, subcutaneous tissue and skin. In the second method the percentage thick reduction of the isolated temporal muscle will be measured and the third the volumetric analysis of the temporal muscle, subcutaneous tissue and skin will be calculated from the superior edge of zygomatic arch to superior temporal line. The functional results wiil be compared using the Modified Rankin Score. Others variables such frontal facial palsy, post-operative hemorrhage, cerebrospinal fistulas, hydrocephalus and mortality will be also analyzed

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of intracranial aneurysms

Exclusion Criteria:

Giant aneurysms Intracranial hematomas

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Atrophy degree measurement (temporal muscle) | 6 months
  The degree of atrophy was measured with three methods. In the first one, the authors observed the percentage of thick reduction in the temporal muscle, subcutaneous tissue and skin. In the second method the percentage thick reduction of the isolated temporal muscle was observed. Both measures were made in the beginning of the sphenoid wing. The volumetric analysis of the temporal muscle, subcutaneous tissue and skin was calculated from the superior edge of zygomatic arch to superior temporal line using the OsiriX software

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo C Welling, MD, Principal Investigator — University of Sao Paulo

REFERENCES:
- [Derived] Welling LC, Figueiredo EG, Wen HT, Gomes MQ, Bor-Seng-Shu E, Casarolli C, Guirado VM, Teixeira MJ. Prospective randomized study comparing clinical, functional, and aesthetic results of minipterional and classic pterional craniotomies. J Neurosurg. 2015 May;122(5):1012-9. doi: 10.3171/2014.11.JNS146. Epub 2014 Dec 19. PMID 25526271